CLINICAL TRIAL: NCT06826001
Title: COMPARISON OF EFFICACY OF TOPICAL FINESTERIDE VERSUS TOPICAL MINOXIDAL IN TREATMENT OF ANDROGENETIC ALOPECIA
Brief Title: Various Procedural Treatment Options for Androgenetic Alopecia
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sheikh Zayed Medical College (Other Government)
Responsible Party: Principal Investigator, Farah Humera, Post Graduate Resident in Dermatology, Sheikh Zayed Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: sheikh-ZMC-FH
Record Dates: First submitted 2025-01-21; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Androgenetic Alopecia
Keywords: androgenetic alopecia; finasteride; minoxidil; hairloss
MeSH Terms: conditions — Alopecia | interventions — Finasteride; Minoxidil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Finesteride group (Active Comparator): Group A will receive topical finasteride spray 0.25% twice daily for 12 weeks
  Interventions: Drug: topical finasteride
- Minoxidil group (Active Comparator): Group B will receive topical 5% minoxidil twice daily for 12 weeks
  Interventions: Drug: Topical minoxidil

INTERVENTIONS:
Drug: topical finasteride — Group A will receive topical finesteride spray 0.25% twice daily for 12 weeks
  Arms: Finesteride group
Drug: Topical minoxidil — Group B will receive topical 5% minoxidal twice daily for 12 weeks
  Arms: Minoxidil group

SUMMARY:
Androgenetic alopecia (AGA)is the most common form of alopecia. It predominantly affects males, but there has been a significant surge in female preponderance too, over the last decade Minoxidil belong to the anti-hypertensive class but it also affects the potassium channels present in vascular smooth muscles and hair follicles. This potassium channel activity may stimulate the microcirculation around the hair follicles and induces arteriolar vasodilation, thereby encouraging conditions conducive to hair growth Topical administration of finasteride offers the potential to reduce systemic effects related to its mechanism of action by preferentially inhibiting 5-a reductase in the scalp, as has been suggested in recent years so in this study we are going to compare efficacy of topical minoxidil versus topical finasteride in treatment of androgenetic alopecia

DETAILED DESCRIPTION:
Androgenetic alopecia (AGA)is considered to be a very common form of alopecia. Minoxidil belong to the anti-hypertensive class but it also affects the potassium channels present in vascular smooth muscles and hair follicles. This potassium channel activity may stimulate the microcirculation around the hair follicles and induces arteriolar vasodilation, thereby encouraging conditions conducive to hair growth The clinical efficacy of oral finasteride for treating AGA is well established. Although oral finasteride is generally well tolerated Topical finasteride is a medication that is used to treat hair loss in men and women. It is a topical version of the oral medication finasteride, which works by blocking the conversion of testosterone to dihydrotestosterone (DHT), a hormone that contributes to hair loss. Topical administration of finasteride offers the potential to reduce systemic effects related to its mechanism of action by preferentially inhibiting 5-a reductase in the scalp, as has been suggested in recent years.

OBJECTIVE "To compare the efficacy of topical finasteride vs topical minoxidil in the treatment of androgenetic alopecia in tertiary care hospital"

DATA COLLECTION:

Data will be collected on prescribed proforma which is attached, at Dermatology OPD, Sheikh Zayed Hospital, Rahim Yar Khan. Patient will be selected on basis of inclusion & exclusion criteria. Informed consent will be taken from selected patients before data collection. Study will include 190 patients which will be divided into 2 groups A & B, 95 in each group. Group A will receive topical finasteride spray 0.25% twice daily for 12 weeks. Group B will receive topical 5% minoxidil twice daily for 12 weeks Patient will be followed at the end of 12 weeks therapy.

DATA ANALYSIS:

Data will be analyzed by SPSS (Statistical Package for the Social Sciences) v25.0.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-50 years
* Gender: Male
* ANDROGENETIC ALOPECIA with AGA stage 2-6 Norwood-Hamilton -classification
* Patients not taking any treatment in last 1 month

Exclusion Criteria:

* Abrasion or abnormalities to the scalp
* Hair transplant
* Hypersensitivity
* Recent history of local infections of the head
* History of relevant significant disease active seborrheic dermatitis
* Concurrent use of :
* corticosteroids
* anabolic steroids or over-the-counter 'hair restorers'
* use of drugs with anti-androgenic properties within 6 months light or laser treatment of the scalp within the last 3 months.

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 190 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
COMPARISON OF EFFICACY OF TOPICAL FINESTERIDE VERSUS TOPICAL MINOXIDAL IN TREATMENT OF ANDROGENETIC ALOPECIA | Clinical assessment for efficacy will be done monthly for 6 months
  The final efficacy will be divided into following groups on the basis of Norwood-Hamilton scale from the baseline :1.Excellent efficacy: It is defined as greater than two scale change in hair density as measured from baseline . 2. moderate efficacy : It is defined as one to two scale change in hair density as measured from baseline. Percentage increase in hair density as clinically measured by the surface area from the baseline. 3.Non efficacious: It is defined as less than one scale change in hair density as measured clinically from baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Sheikh zayed Medical College and Hospital, Rahim Yar Khan, Punjab 644200, Rahim Yar Khan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No